CLINICAL TRIAL: NCT00002502
Title: BUSULFAN AND CYCLOPHOSPHAMIDE FOR CYTOREDUCTION OF PATIENTS WITH ACUTE AND CHRONIC LEUKEMIAS AND MYELODYSPLASTIC SYNDROMES UNDERGOING ALLOGENEIC BONE MARROW TRANSPLANTATION WHO CANNOT BE TREATED WITH TOTAL BODY IRRADIATION
Brief Title: Combination Chemotherapy and Bone Marrow Transplantation in Treating Patients With Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 92-103; CDR0000077927 (Registry Identifier: PDQ (Physician Data Query)); NCI-H92-0143
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; childhood Burkitt lymphoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; chronic myelomonocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; intraocular lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Busulfan; Cyclophosphamide; Cytarabine

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of busulfan and cyclophosphamide followed by bone marrow transplantation in treating patients who have acute or chronic leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of marrow ablation with high dose busulfan/cyclophosphamide on engraftment, incidence of posttransplant relapse, incidence and severity of graft versus host disease (GVHD), and incidence and severity of nonGVHD posttransplant complications in patients with acute or chronic leukemia or myelodysplastic syndrome who are eligible for allogeneic bone marrow transplants from HLA identical/compatible donors but who cannot or should not receive total body irradiation as part of their cytoreductive regimen.

OUTLINE: 2-Drug Combination Cytoreductive Chemotherapy followed by Bone Marrow Transplant with, as indicated, CNS Prophylaxis. Busulfan, BU, NSC-750; Cyclophosphamide, CTX, NSC-26271; followed by Allogeneic Bone Marrow, AlBM; with, as indicated, Intrathecal Cytarabine, IT ARA-C, NSC-63878.

PROJECTED ACCRUAL: At least 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary or secondary acute nonlymphocytic leukemia and acute lymphocytic leukemia in one of the following states: First or greater remission Early relapse Chronic myelogenous leukemia (CML) in one of the following states: First or greater chronic phase Treatment on this protocol is preferred to total body irradiation containing protocols for patients under 40 with CML in stable first chronic phase who are otherwise eligible for allogeneic bone marrow transplantation Accelerated phase Myeloid or lymphoid blast crisis Myelodysplastic syndromes of the following types: Refractory anemia Refractory anemia with ringed sideroblasts Refractory anemia with excess blasts Chronic myelomonocytic leukemia Multiple myeloma Non-Hodgkin's lymphoma HLA identical bone marrow donor available Unable to undergo total body irradiation because of one of the following reasons: Under age 2 (CNS still growing and at high risk of permanent radiation injury) Prior high dose radiotherapy to the brain, lungs, heart, liver, or abdomen In relapse following allogeneic or autologous transplant using total body irradiation for ablation, but eligible for a second transplant No current CNS involvement

PATIENT CHARACTERISTICS: Age: 50 and under (patients aged 51-55 accrued on a case-by-case basis after discussion and approval by the BMT service) Performance status: Karnofsky 70-100% Life expectancy: Greater than 8 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 mg/dL AST no greater than 3 times normal Neither value increasing for at least 2-4 weeks prior to transplant Renal: Creatinine less than 2 times normal and not rising for at least 2-4 weeks prior to transplant OR Creatinine clearance greater than 80 mL/min Cardiovascular: Left ventricular ejection fraction at least 50% Cardiac function good Pulmonary: No severe restrictive lung disease No chronic obstructive pulmonary disease Other: No active viral or bacterial infection at transplant No coexisting medical problem that would significantly increase the risk of the transplant procedure Not pregnant

PRIOR CONCURRENT THERAPY: Prior therapy allowed, including prior bone marrow transplant

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1992-07; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza B. Papadopoulos, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States